CLINICAL TRIAL: NCT00731627
Title: Simvastatin in Aneurysmal Subarachnoid Haemorrhage (STASH) a Multicentre Randomised Controlled Clinical Trial
Acronym: STASH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Mr PJ Kirkpatrick, Consultant Neurosurgeon, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-000277-30; ISRCTN75948817
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Subarachnoid Haemorrhage
Keywords: intracranial aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): placebo
  Interventions: Drug: placebo
- 11 (Active Comparator): simvastatin
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: placebo — one tablet a day for up to 21 days
  Other Names: placebo tablet
  Arms: 1
Drug: simvastatin — simvastatin 40mg once a day for a maximum of 21 days
  Other Names: ritechol
  Arms: 11

SUMMARY:
Intracranial bleeding from ruptured blood vessels (called a subarachnoid haemorrhage -SAH) affects 7000 patients each year in the UK and is a source of considerable death and disability, even in young adults. Recent observations indicate that these bleeds can cause reduced cerebral blood flow which leads to a bad outcome. High rates of death and disability occur, and are particularly prevalent when low cerebral blood flow results in stroke. Prevention of cerebral artery spasm and improvement in blood vessel reflexes are the target of modern therapy. Candidate drugs include statins which have an impeccable safety record and multiple potential beneficial actions (improve cerebral blood flow, reduce inflammatory processes, reduce adverse blood coagulation) following SAH.

The investigators plan to use a statin, Simvastatin (40 mg) to improve cerebral blood flow and reduce inflammation. We have already completed a phase 11 study (n=80) which demonstrated potential benefits for acute statin therapy following SAH, and the investigators now wish to conduct a multi-centre phase 111 study to explore any potential clinical benefits in a larger population (n=1600). The purpose is to see whether the positive effects of statins seen in our phase II study translate into clinical benefits - both short term (e.g. reduced need for intensive care) and long term (outcome and wellbeing at 6 months).

ELIGIBILITY:
Inclusion Criteria

* Patients (age 18 - 65 yr) in which the admitting neurosurgeon has confirmatory evidence of an aneurysm, either by CT angiography, MR angiography or DSA.
* Any clinical grade accepted provided a reasonable prospect of survival.
* Delay to randomisation and initiation of trial medication from the time of the presenting ictus does not exceed 96 hours.

Exclusion Criteria

* Unsalvageable patients:Fixed and dilated pupils after resuscitation, and/or a devastating scan, which precludes definitive therapy.
* Already taking statin therapy.
* Those taking Warfarin - type drugs.
* Pregnancy.
* Known renal or hepatic impairment
* Suspected or known additional disease process, which threatens life expectancy (e.g.malignancy).
* Known or strong suspicion of drug abuse, alcoholism, or those who are unlikely to be amenable to 6 month follow up.
* Those already taking amiodarone, verapamil or potent CYP3A4 inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2007-01; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Disability Score (mRS) at 6 months | 6-12 months

SECONDARY OUTCOMES:
Need and intensity of delayed ischaemic deficit rescue therapy | 1-3 months
Incidence and duration of delayed ischaemic deficits | 1-3 months
Incidence and severity of sepsis | 1-3 months
Length of intensive care and total acute hospital stay | 1-3 months
Discharge destination | 1-3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dept of Neurological Surgery, University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida

REFERENCES:
- [Derived] Budohoski KP, Czosnyka M, Kirkpatrick PJ. The Role of Monitoring Cerebral Autoregulation After Subarachnoid Hemorrhage. Neurosurgery. 2015 Aug;62 Suppl 1:180-4. doi: 10.1227/NEU.0000000000000808. No abstract available. PMID 26181941